CLINICAL TRIAL: NCT04542499
Title: A Phase 3, Double-Blind, Randomized, Placebo-Controlled, Parallel-Group, Flexible-Dose, 27-Week Trial to Evaluate the Efficacy, Safety, and Tolerability of Tavapadon as Adjunctive Therapy for Parkinson's Disease in Levodopa-Treated Adults With Motor Fluctuations (TEMPO-3 Trial)
Brief Title: Flexible-Dose, Adjunctive Therapy Trial in Adults With Parkinson's Disease With Motor Fluctuations (TEMPO-3)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CVL-751-PD-003; 2019-002951-40 (EudraCT Number)
Record Dates: First submitted 2020-09-02; First posted 2020-09-09 (Actual); Results first posted 2025-03-25 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Parkinson Disease
Keywords: Parkinsonian Disorders; Brain Diseases; Central Nervous System Diseases; Nervous System Disease; Movement Disorders; Neurodegenerative Diseases
MeSH Terms: conditions — Parkinson Disease; Parkinsonian Disorders; Brain Diseases; Central Nervous System Diseases; Nervous System Diseases; Movement Disorders; Neurodegenerative Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Tavapadon (Experimental): Participants will receive a tavapadon tablet titrated 5 to 15milligrams (mg) once daily (QD)orally for 27 weeks.
  Interventions: Drug: Tavapadon
- Placebo (Placebo Comparator): Participants will receive placebo matching to tavapadon tablet QD orally for 27 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tavapadon — Participants will be randomized to receive tavapadon 5 to 15 mg tablet QD orally for 27 weeks.
  Other Names: PF-06649751; CVL-751
  Arms: Tavapadon
Drug: Placebo — Participants will receive placebo matching to tavapadon QD orally for 27 weeks.
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the effect of tavapadon on the change from baseline in total daily hours of "on" time without troublesome dyskinesia in L-Dopa-treated participants with Parkinson's Disease (PD) who are experiencing motor fluctuations.

ELIGIBILITY:
Key Inclusion Criteria:

* Male and female participants aged 40 to 80 years, inclusive, at the time of signing the informed consent form (ICF).
* Sexually active men or women of childbearing potential must agree to use acceptable (at minimum) or highly effective birth control, or remain abstinent during the trial and for 4 weeks after the last dose of trial treatment.
* Participants who are capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the ICF and in this protocol.
* Participants with a diagnosis of PD that is consistent with the UK Parkinson's Disease Society Brain Bank diagnostic criteria, with bradykinesia and motor asymmetry.
* Participants with modified Hoehn and Yahr stage 2, 2.5, or 3 in the "on" state.
* Participants with a good response to levodopa (L- Dopa) in the judgment of the investigator.
* Participants who return a completed self-reported home diary for motor function status (Hauser diary) during the screening period (after diary training and concordance testing has occurred), with recordings for 2 consecutive days (ie, 2 consecutive 24-hour periods) showing at least 2 and half hours of "off" time on each of the 2 days.
* Participants who are on a stable dose of L-Dopa for at least 4 weeks prior to screening and are taking a minimum total daily dose of 400 milligram (mg) divided in at least 4 doses per day of standard carbidopa/levodopa or divided in at least 3 doses per day of extended-release carbidopa/levodopa capsules. The carbidopa/levodopa dose and frequency must be maintained for the duration of the trial.
* Prior and concurrent use of catechol-O-methyltransferase (COMT) inhibitors, monoamine oxidaseB (MAO-B) inhibitors, amantadine, istradefylline or anticholinergic drugs are permitted if the use was initiated greater than (>) 90 days before the baseline visit and the dosage will remain stable for the duration of the trial (ie, no change in the COMT,MAO-B inhibitor, amantadine, istradefylline or anticholinergic dose is permitted during the trial).

Key Exclusion Criteria:

* Participants with a history or clinical features consistent with essential tremor, atypical or secondary parkinsonian syndrome (including, but not limited to, progressive supranuclear palsy, multiple system atrophy, cortico-basal degeneration, or drug-induced or post stroke parkinsonism).
* Participants with a history of nonresponse or insufficient response to L-Dopa at therapeutic dosages.
* Participants with a history or current diagnosis of a clinically significant impulse control disorder(Disruptive, Impulse Control, and Conduct Disorder per DSM-5).
* Participants with the presence of or history of brain tumor, hospitalization for severe head trauma, epilepsy (as defined by the International League Against Epilepsy), or seizures.
* Participants with a history of psychosis or hallucinations within the previous 12 months.
* Participants who answer "yes" on the Columbia-Suicide Severity Rating Scale (C-SSRS) Suicidal Ideation Item 4 or Item 5 (Active Suicidal Ideation with Some Intent to Act, Without Specific Plan, or Active Suicidal Ideation with Specific Plan and Intent)and whose most recent episode meeting the criteria for C-SSRS Item 4 or Item 5 occurred within the last6 months, OR Participants who answer "yes" on any of the 5 C-SSRS Suicidal Behavior Items (actual attempt, interrupted attempt, aborted attempt, preparatory acts, or behavior) and whose most recent episode meeting the criteria for any of these 5C-SSRS Suicidal Behavior Items occurred within the last 2 years, OR Participants who, in the opinion of the investigator, present a serious risk of suicide.
* Participants with substance abuse or dependence disorder, including alcohol, benzodiazepines, and opioids, but excluding nicotine, within the past 6months (180 days).
* Participants with dementia or cognitive impairment that, in the judgement of the investigator, would exclude the participant from understanding the ICF or participating in the trial.
* Participants with any condition that could possibly affect drug absorption, including bowel resections, bariatric weight loss surgery, or gastrectomy (this does not include gastric banding).
* Participants who have a positive result for human immunodeficiency virus (HIV) antibodies, hepatitis B surface antigen (HbsAg), or hepatitis C virus (HCV)antibodies at screening.
* Participants with a history of myocardial infarction with residual atrial, nodal, or ventricular arrhythmias that are not controlled with medical and/or surgical intervention; second- or third-degree atrioventricular block; sick sinus syndrome; severe or unstable angina; or congestive heart failure within the last 12months. A recent (less than or equal to [<=12]months) history of myocardial infarction with secondary arrhythmias is exclusionary regardless of the therapeutic control.
* Participants with a history of neuroleptic malignant syndrome.
* Participants who are currently receiving moderate or strong CYP3A4 inducers or CYP3A4 inhibitors(except for topical administration).
* Participants with a positive urine drug screen for illicit drugs are excluded and may not be retested or rescreened. Participants with a positive urine drug screen resulting from use of marijuana (any tetrahydrocannabinol-containing product),prescription, or over-the-counter medications or products that, in the investigator's documented opinion, do not signal a clinical condition that would impact the safety of the participant or interpretation of the trial results may continue evaluation for the trial following consultation and approval by the medical monitor
* Participants with a Montreal Cognitive Assessment(MoCA) score <26.
* Participants with clinically significant orthostatic hypotension (eg, syncope).
* Participants with a 12-lead ECG demonstrating aQTcF interval >450 msec.
* Participants with moderate or severe renal impairment (creatinine clearance as estimated by Cockcroft-Gault formula <30 mL/min or on dialysis).
* Participants with any of the following abnormalities in clinical laboratory tests at the Screening Visit, as assessed by the central laboratory and confirmed by a single repeat measurement, if deemed necessary:
* Aspartate Aminotransferase (AST) or Alanine Aminotransferase (ALT) >=3 × Upper Limit Normal (ULN).
* Total bilirubin >=1.5 × ULN. Participants with a history of Gilbert's syndrome may be eligible provided they have a value <ULN for direct bilirubin
* Participants with other abnormal laboratory test results, vital sign results, or ECG findings unless, in the judgment of the investigator, the findings are not medically significant and would not impact the safety of the participants or the interpretation of the trial results.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 507 (Actual)
Dates: Start 2020-09-23 (Actual); Primary Completion 2024-01-29 (Actual); Study Completion 2024-02-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (134):
- United States (51):
  - Pheonix, Arizona, Phoenix, Arizona
  - Little Rock, Arkansas, Little Rock, Arkansas
  - Fountain Valley, California, Fountain Valley, California
  - Fresno, California, Fresno, California
  - Long beach, California, Long Beach, California
  - Los Angeles, California, Los Angeles, California
  - Pasadena, California, Pasadena, California
  - Reseda, California, Reseda, California
  - Denver, Colorado, Denver, Colorado
  - Englewood, Colorado, Englewood, Colorado
  - Adventura, Florida, Adventura, Florida
  - Atlantis, Florida, Atlantis, Florida
  - Boca Raton, Florida, Boca Raton, Florida
  - Coral Springs, Florida, Coral Springs, Florida
  - Hallandale Beach, Florida, Hallandale, Florida
  - Maitland, Florida, Maitland, Florida
  - Ocala, Florida, Ocala, Florida
  - Port Charlotte, Florida, Port Charlotte, Florida
  - Port Orange, Florida, Port Orange, Florida
  - Tampa, Florida, Tampa, Florida
  - Winter Park, Florida, Winter Park, Florida
  - Augusta, Georgia, Augusta, Georgia
  - Chicago, Illinois, Chicago, Illinois
  - Elk Grove Village, Illinois, Elk Grove Village, Illinois
  - Kansas City, Kansas, Kansas City, Kansas
  - Lexington, Kentucky, Lexington, Kentucky
  - Scarborough, Maine, Scarborough, Maine
  - Boston, Massachusettes, Boston, Massachusetts
  - Boston Neuro Research Center, North Dartmouth, Massachusetts
  - Farmington Hills, Michigan, Farmington Hills, Michigan
  - West Bloomfield, Michigan, West Bloomfield, Michigan
  - Saint Louis, Missouri, St Louis, Missouri
  - Las Vegas, Nevada, Las Vegas, Nevada
  - Syracuse, New York, Syracuse, New York
  - Asheville, North Carolina, Asheville, North Carolina
  - Cincinnati, Ohio, Cincinnati, Ohio
  - Cleveland, Ohio, Cleveland, Ohio
  - Columbus, Ohio, Columbus, Ohio
  - Dayton, Ohio, Dayton, Ohio
  - Toledo, Ohio, Toledo, Ohio
  - Memphis, Tennessee, Memphis, Tennessee
  - Cypress, Texas, Cypress, Texas
  - Georgetown, Texas, Georgetown, Texas
  - Houston, Texas, Houston, Texas
  - Lubbock, Texas, Lubbock, Texas
  - Round Rock, Texas, Round Rock, Texas
  - Burlington, Vermont, Burlington, Vermont
  - Richmond, Virginia, Richmond, Virginia
  - Virginia Beach, Virginia, Virginia Beach, Virginia
  - Kirkland, Washington, Kirkland, Washington
  - Spokane, Washington, Spokane, Washington
- Australia (5):
  - Clayton VIC, Clayton, Clayton VIC
  - Erina, New South Wales, Erina, New South Wales
  - Kogarah, New South Wales, Kogarah, New South Wales
  - Woolloongabba, Queensland, Woolloongabba, Queensland
  - Parkville, Victoria, Parkville, Victoria
- Bulgaria (5):
  - Pleven, Bulgaria, Pleven
  - Pleven, Pleven
  - Multiprofile Hospital, Sofia, Sofia
  - Sofia, Sofia
  - DCC Neoclinic, Sofia
- Canada (2):
  - Ottawa, Ontario, Ottawa, Ontario
  - Toronto, Ontario, Toronto, Ontario
- Czechia (4):
  - Chocen, Choceň, Chocen
  - Prague, Czech Republic, Prague, Czech Republic
  - Prague,, Prague
  - Rychnov nad Kněžnou, Rychnov nad Kněžnou
- France (6):
  - Creteil,, Créteil, Creteil
  - Boulevard Pinel, Bron, Bron
  - Nantes CEDEX 1, Nantes
  - Nîmes cedex, Nîmes
  - Strasbourg, Strasbourg
  - Toulouse Cedex 9, Toulouse
- Germany (11):
  - Muenster, Münster, Muenster
  - Bad Homburg, Bad Homburg
  - Berlin, Berlin
  - Bochum, Bochum
  - Brandenburg, Germany, Brandenburg
  - Duesseldorf,, Düsseldorf
  - Gera, Gera
  - Haag in Oberbayern, Haag in Oberbayern
  - Klinikum rechts der Isar der TU München, Munich
  - Muenchen, München
  - Stadtroda, Stadtroda
- Hungary (4):
  - Gyor,, Győr, Gyor
  - Budapest, Budapest
  - Pecs, Pécs
  - Szeged, Szeged
- Israel (6):
  - Ashkelon, Ashkelon
  - Haifa, Haifa
  - Jerusalem, Jerusalem
  - Petah Tiqva, Petah Tikva
  - Shoham, Shoham
  - Tel Aviv, Tel Aviv
- Italy (8):
  - Ancona, Ancona
  - Cassino, Cassino
  - Milano, Milan
  - Padova, Padua
  - Pisa, Pisa
  - Rome, Rome
  - Rozzano Milano, Rozzano
  - Torino, Torino
- Poland (12):
  - Cracow, Krakow, Cracow
  - Krakow, Krakow, Krakow
  - Bydgoszcz, Kujawsko-Pomorskie, Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Siemianowice Slaskie, Siemianowice Śląskie, Siemianowice Slaskie
  - Katowice, Katowice
  - Kraków, Krakow
  - Krakow, Krakow
  - Lublin, Lublin
  - Centrum Medyczne Hope Clinic Sebastian Szklener, Lublin
  - Warsaw, Warsaw
  - Singua, Warsaw
  - Lodz, Lodz, Łódź Voivodeship
- Serbia (4):
  - Belgrade, Serbia, Belgrade
  - Belgrade,, Belgrade
  - Belgrade, Belgrade
  - Belgrade, Kragujevac, Belgrade
- Spain (9):
  - Elche, Elche, Alicante
  - Barcelona, Barcelona
  - San Sebastian, Donostia / San Sebastian
  - Madrid, Madrid
  - Madrid, Spain, Madrid
  - Pamplona, Pamplona
  - Sevilla, Seville
  - Terrassa, Terrassa
  - Valencia, Valencia
- Ukraine (7):
  - Zaporiizhzhya, Zaporizhzhya, Zaporiizhzhya
  - Zaporozhya, Zaporizhzhya, Zaporozhya
  - Dnipro, Dnipro
  - Kharkiv, Kharkiv
  - Kiev, Kiev
  - Lviv, Lviv
  - Vinnitsa, Vinnitsa

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=CVL-751-PD-003

RESULTS

PARTICIPANT FLOW:
Recruitment Details: In this Phase 3, Double-Blind study, a total of 368 subjects with Parkinson's Disease(PD) were be randomized in a 1:1 ratio to receive Tavapadon (5 mg to 15 mg) or Placebo once daily (QD) for 27 Weeks.
Period: Overall Study
Arm/Group | Placebo | Tavapadon
Started | 255 | 252
Completed | 206 | 159
Not Completed | 49 | 93
Not completed — Adverse Event | 23 | 43
Not completed — Lack of Efficacy | 5 | 2
Not completed — Lost to Follow-up | 3 | 4
Not completed — Failure to Meet Continuation Criteria | 0 | 1
Not completed — Treatment with Prohibited Concomitant Medications | 1 | 0
Not completed — Non-Compliance with Study Drug | 0 | 2
Not completed — Physician Decision | 0 | 1
Not completed — Site Terminated by Sponsor | 3 | 5
Not completed — Withdrawal by Subject | 12 | 33
Not completed — Other | 2 | 2

BASELINE CHARACTERISTICS:
Population: Includes all enrolled subjects that received at least one dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Tavapadon | Total
Number analyzed (Participants) | 255 | 252 | 507
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.1 (8.52) | 65.6 (8.42) | 64.9 (8.49)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 85 | 101 | 186
  Male | 170 | 151 | 321
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 16 | 11 | 27
  Not Hispanic or Latino | 232 | 226 | 458
  Unknown or Not Reported | 7 | 15 | 22
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 2
  Asian | 2 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 2 | 6
  White | 245 | 246 | 491
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 2 | 4
ON Time (hours) Without Troublesome Dyskinesia at Baseline [Mean (Standard Deviation); unit: hours] — Population: Population includes subjects who received at least one dose of study drug and had available data for analysis.
  hours
    number analyzed (Participants) | 248 | 247 | 495
    (all) | 10.148 (2.637) | 9.884 (2.569) | 10.016 (2.604)
OFF Time (hours) at Baseline [Mean (Standard Deviation); unit: hours] — Population: Population includes subjects who received at least one dose of study drug and had available data for analysis.
  hours
    number analyzed (Participants) | 248 | 247 | 495
    (all) | 5.408 (2.484) | 5.638 (2.246) | 5.523 (2.369)
Movement Disorder Society - Unified Parkinson's Disease Rating Score at Baseline (Parts I, II, III) [Mean (Standard Deviation); unit: units on a scale] — The MDS-UPDRS rating tool was used to follow longitudinal course of Parkinson's Disease. It was made up of 4 parts: Part 1: Non-motor aspects of experiences of daily living (13 items. Score range: 0-52); Part 2: Motor aspects of experiences of daily living (13 items. Score range: 0-52); Part 3: Motor examination (18 items. Score range: 0-132); Part 4: Motor complications (6 items. Score range: 0-24. Part 4 was not collected in this trial). Each item has 0-4 rating on scale from 0 (normal) to 4 (severe). Higher values represent a worse outcome.
  units on a scale
    Part I | 7.5 (4.93) | 8.0 (5.13) | 7.7 (5.03)
    Part II | 12.5 (7.05) | 13.3 (6.54) | 12.9 (6.80)
    Part III | 32.4 (14.26) | 32.6 (14.34) | 32.5 (14.29)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Total "On" Time Without Troublesome Dyskinesia Based on the 2-day Average of the Self-completed Home Diary for Motor Function Status (Hauser Diary)
Description: The Hauser diary assesses participant-defined clinical status over a period of time and provides a tool for assessment of the change in "off" time and "on" time with troublesome dyskinesia (which is a more accurate reflection of clinical response than "off" time alone). The Hauser diary asks participants to rate their mobility for each 30-minute period and to record their status for the majority of the period in 1 of 5 categories as: "on" time without dyskinesia, "on" time with nontroublesome dyskinesia, "on" time with troublesome dyskinesia, "off" time, or asleep. The total "on" time without troublesome dyskinesia will be assessed and reported at endpoint.
Time Frame: Week 26
Population: Population includes subjects who received at least one dose of study drug and had available data for analysis.
Measure: Least Squares Mean (Standard Error); unit: hours
Arm/Group | Placebo | Tavapadon
Number analyzed (Participants) | 201 | 153
hours | 0.619 (0.188) | 1.721 (0.207)
Statistical Analysis 1: Comparison: Placebo vs Tavapadon; Test type: Superiority; p < 0.0001, Mixed-effect Model Repeated Measurement — LS Means, SE, difference from placebo, and confidence intervals are estimated using a mixed effects repeated measures model with fixed effects for treatment group, visits, and treatment by visit interaction and baseline as a covariate; LS Mean of Difference = 1.103, 95% CI 2-sided [0.553 to 1.653], Standard Error of Mean 0.280

2. Secondary Outcome: Change From Baseline in Total Daily "Off" Time Based on the 2-Day Average of the Self-Completed Home Diary for Motor Function Status (Hauser Diary)
Description: The Hauser diary assesses participant-defined clinical status over a period of time and provides a tool for assessment of the change in "off" time and "on" time with troublesome dyskinesia (which is a more accurate reflection of clinical response than "off" time alone). The Hauser diary asks participants to rate their mobility for each 30-minute period and to record their status for the majority of the period in 1 of 5 categories as: "on" time without dyskinesia, "on" time with nontroublesome dyskinesia, "on" time with troublesome dyskinesia, "off" time, or asleep. The total daily "Off" time will be assessed and reported at endpoint.
Time Frame: Week 26
Population: Population includes subjects who received at least one dose of study drug and had available data for analysis.
Measure: Least Squares Mean (Standard Error); unit: hours
Arm/Group | Placebo | Tavapadon
Number analyzed (Participants) | 201 | 153
hours | -0.933 (0.182) | -1.876 (0.200)
Statistical Analysis 1: Comparison: Placebo vs Tavapadon; Test type: Superiority; p = 0.0006, Mixed-effect Model Repeated Measurement — [p-value comment as in outcome 1, analysis 1]; LS Mean of Difference = -0.943, 95% CI 2-sided [-1.475 to -0.410], Standard Error of Mean 0.271

3. Secondary Outcome: Change From Baseline in the Total "On" Time Without Troublesome Dyskinesia Based on the 2-day Average of the Self-completed Home Diary for Motor Function Status (Hauser Diary)
Description: The Hauser diary assesses participant-defined clinical status over a period of time and provides a tool for assessment of the change in "off" time and "on" time with troublesome dyskinesia (which is a more accurate reflection of clinical response than "off" time alone). The Hauser diary asks participants to rate their mobility for each 30-minute period and to record their status for the majority of the period in 1 of 5 categories as: "on" time without dyskinesia, "on" time with nontroublesome dyskinesia, "on" time with troublesome dyskinesia, "off" time, or asleep. The total "on" time without troublesome dyskinesia will be assessed and reported at different time points.
Time Frame: Week 2, 5, 8, 11, 14, 18, 22, and 26
Population: Population includes subjects who received at least one dose of study drug and had available data for analysis.
Measure: Least Squares Mean (Standard Error); unit: hours
Arm/Group | Placebo | Tavapadon
Number analyzed (Participants) | 245 | 242
hours
  Week 2: number analyzed (Participants) | 239 | 239
  Week 2 | 0.535 (0.133) | 0.305 (0.133)
  Week 5: number analyzed (Participants) | 234 | 223
  Week 5 | 0.516 (0.148) | 0.616 (0.151)
  Week 8: number analyzed (Participants) | 229 | 206
  Week 8 | 0.470 (0.162) | 1.052 (0.168)
  Week 11: number analyzed (Participants) | 218 | 192
  Week 11 | 0.705 (0.163) | 1.063 (0.171)
  Week 14: number analyzed (Participants) | 218 | 182
  Week 14 | 0.584 (0.175) | 1.282 (0.187)
  Week 18: number analyzed (Participants) | 206 | 174
  Week 18 | 0.623 (0.174) | 1.592 (0.185)
  Week 22: number analyzed (Participants) | 202 | 163
  Week 22 | 0.870 (0.177) | 1.749 (0.190)
  Week 26: number analyzed (Participants) | 201 | 153
  Week 26 | 0.619 (0.188) | 1.721 (0.207)
Statistical Analysis 1: Comparison: Placebo vs Tavapadon; Week 2; Test type: Superiority; p = 0.2216, Mixed-effect Model Repeated Measurement — [p-value comment as in outcome 1, analysis 1]; LS Mean of Difference = -0.230, 95% CI 2-sided [-0.600 to 0.139], Standard Error of Mean 0.188
Statistical Analysis 2: Comparison: Placebo vs Tavapadon; Week 5; Test type: Superiority; p = 0.6379, Mixed-effect Model Repeated Measurement — [p-value comment as in outcome 1, analysis 1]; LS Mean of Difference = 0.099, 95% CI 2-sided [-0.316 to 0.515], Standard Error of Mean 0.211
Statistical Analysis 3: Comparison: Placebo vs Tavapadon; Week 8; Test type: Superiority; p = 0.0132, Mixed-effect Model Repeated Measurement — [p-value comment as in outcome 1, analysis 1]; LS Mean of Difference = 0.582, 95% CI 2-sided [0.122 to 1.042], Standard Error of Mean 0.234
Statistical Analysis 4: Comparison: Placebo vs Tavapadon; Week 11; Test type: Superiority; p = 0.1299, Mixed-effect Model Repeated Measurement — [p-value comment as in outcome 1, analysis 1]; LS Mean of Difference = 0.358, 95% CI 2-sided [-0.106 to 0.821], Standard Error of Mean 0.236
Statistical Analysis 5: Comparison: Placebo vs Tavapadon; Week 14; Test type: Superiority; p = 0.0068, Mixed-effect Model Repeated Measurement — [p-value comment as in outcome 1, analysis 1]; LS Mean of Difference = 0.698, 95% CI 2-sided [0.194 to 1.202], Standard Error of Mean 0.257
Statistical Analysis 6: Comparison: Placebo vs Tavapadon; Week 18; Test type: Superiority; p = 0.0002, Mixed-effect Model Repeated Measurement — [p-value comment as in outcome 1, analysis 1]; LS Mean of Difference = 0.969, 95% CI 2-sided [0.469 to 1.469], Standard Error of Mean 0.254
Statistical Analysis 7: Comparison: Placebo vs Tavapadon; Week 22; Test type: Superiority; p = 0.0008, Mixed-effect Model Repeated Measurement — [p-value comment as in outcome 1, analysis 1]; LS Mean of Difference = 0.879, 95% CI 2-sided [0.369 to 1.389], Standard Error of Mean 0.259
Statistical Analysis 8: Comparison: Placebo vs Tavapadon; Week 26; Test type: Superiority; p < 0.0001, Mixed-effect Model Repeated Measurement — [p-value comment as in outcome 1, analysis 1]; LS Mean of Difference = 1.103, 95% CI 2-sided [0.553 to 1.653], Standard Error of Mean 0.280

4. Secondary Outcome: Change From Baseline in Total Daily "Off" Time Based on the 2-Day Average of the Self-Completed Home Diary for Motor Function Status (Hauser Diary)
Description: The Hauser diary assesses participant-defined clinical status over a period of time and provides a tool for assessment of the change in "off" time and "on" time with troublesome dyskinesia (which is a more accurate reflection of clinical response than "off" time alone). The Hauser diary asks participants to rate their mobility for each 30-minute period and to record their status for the majority of the period in 1 of 5 categories as: "on" time without dyskinesia, "on" time with nontroublesome dyskinesia, "on" time with troublesome dyskinesia, "off" time, or asleep. The total daily "Off" time will be assessed and reported at different time points.
Time Frame: Week 2, 5, 8, 11, 14, 18, 22, and 26
Population: Population includes subjects who received at least one dose of study drug and had available data for analysis.
Measure: Least Squares Mean (Standard Error); unit: hours
Arm/Group | Placebo | Tavapadon
Number analyzed (Participants) | 245 | 242
hours
  Week 2: number analyzed (Participants) | 239 | 239
  Week 2 | -0.598 (0.127) | -0.490 (0.127)
  Week 5: number analyzed (Participants) | 234 | 223
  Week 5 | -0.612 (0.144) | -0.849 (0.146)
  Week 8: number analyzed (Participants) | 229 | 206
  Week 8 | -0.549 (0.153) | -1.367 (0.159)
  Week 11: number analyzed (Participants) | 218 | 192
  Week 11 | -0.876 (0.156) | -1.629 (0.164)
  Week 14: number analyzed (Participants) | 218 | 182
  Week 14 | -0.779 (0.173) | -1.682 (0.185)
  Week 18: number analyzed (Participants) | 206 | 174
  Week 18 | -0.786 (0.176) | -1.810 (0.187)
  Week 22: number analyzed (Participants) | 202 | 163
  Week 22 | -1.014 (0.179) | -1.993 (0.191)
  Week 26: number analyzed (Participants) | 201 | 153
  Week 26 | -0.933 (0.182) | -1.876 (0.200)
Statistical Analysis 1: Comparison: Placebo vs Tavapadon; Week 2; Test type: Superiority; p = 0.5471, Mixed-effect Model Repeated Measurement — [p-value comment as in outcome 1, analysis 1]; LS Mean of Difference = 0.108, 95% CI 2-sided [-0.245 to 0.461], Standard Error of Mean 0.180
Statistical Analysis 2: Comparison: Placebo vs Tavapadon; Week 5; Test type: Superiority; p = 0.2488, Mixed-effect Model Repeated Measurement — [p-value comment as in outcome 1, analysis 1]; LS Mean of Difference = -0.237, 95% CI 2-sided [-0.640 to 0.166], Standard Error of Mean 0.205
Statistical Analysis 3: Comparison: Placebo vs Tavapadon; Week 8; Test type: Superiority; p = 0.0002, Mixed-effect Model Repeated Measurement — [p-value comment as in outcome 1, analysis 1]; LS Mean of Difference = -0.818, 95% CI 2-sided [-1.252 to -0.384], Standard Error of Mean 0.221
Statistical Analysis 4: Comparison: Placebo vs Tavapadon; Week 11; Test type: Superiority; p = 0.0010, Mixed-effect Model Repeated Measurement — [p-value comment as in outcome 1, analysis 1]; LS Mean of Difference = -0.753, 95% CI 2-sided [-1.199 to -0.307], Standard Error of Mean 0.227
Statistical Analysis 5: Comparison: Placebo vs Tavapadon; Week 14; Test type: Superiority; p = 0.0004, Mixed-effect Model Repeated Measurement — [p-value comment as in outcome 1, analysis 1]; LS Mean of Difference = -0.904, 95% CI 2-sided [-1.403 to -0.405], Standard Error of Mean 0.254
Statistical Analysis 6: Comparison: Placebo vs Tavapadon; Week 18; Test type: Superiority; p < 0.0001, Mixed-effect Model Repeated Measurement — [p-value comment as in outcome 1, analysis 1]; LS Mean of Difference = -1.024, 95% CI 2-sided [-1.528 to -0.520], Standard Error of Mean 0.256
Statistical Analysis 7: Comparison: Placebo vs Tavapadon; Week 22; Test type: Superiority; p = 0.0002, Mixed-effect Model Repeated Measurement — [p-value comment as in outcome 1, analysis 1]; LS Mean of Difference = -0.979, 95% CI 2-sided [-1.493 to -0.465], Standard Error of Mean 0.261
Statistical Analysis 8: Comparison: Placebo vs Tavapadon; Week 26; Test type: Superiority; p = 0.0006, Mixed-effect Model Repeated Measurement — [p-value comment as in outcome 1, analysis 1]; LS Mean of Difference = -0.943, 95% CI 2-sided [-1.475 to -0.410], Standard Error of Mean 0.271

5. Secondary Outcome: Change From Baseline in the Movement Disorder Society - Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Parts I, II and III Individual Score
Description: The MDS-UPDRS rating tool was used to follow longitudinal course of Parkinson's Disease. It was made up of 4 parts: Part 1: Non-motor aspects of experiences of daily living (13 items. Score range: 0-52); Part 2: Motor aspects of experiences of daily living (13 items. Score range: 0-52); Part 3: Motor examination (18 items. Score range: 0-132); Part 4: Motor complications (6 items. Score range: 0-24. Part 4 was not collected in this trial). Each item has 0-4 rating on scale from 0 (normal) to 4 (severe). Higher values represent a worse outcome.
Time Frame: Week 26
Population: Population includes subjects who received at least one dose of study drug and had available data for analysis.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Tavapadon
Number analyzed (Participants) | 245 | 242
units on a scale
  Part I: number analyzed (Participants) | 200 | 156
  Part I | 0.0 (0.27) | 0.4 (0.30)
  Part II: number analyzed (Participants) | 200 | 156
  Part II | -0.1 (0.35) | -1.4 (0.39)
  Part III: number analyzed (Participants) | 199 | 156
  Part III | -4.6 (0.65) | -7.0 (0.71)
Statistical Analysis 1: Comparison: Placebo vs Tavapadon; Part I; Test type: Superiority; p = 0.3265, Mixed-effect Model Repeated Measurement — [p-value comment as in outcome 1, analysis 1]; LS Mean of Difference = 0.4, 95% CI 2-sided [-0.4 to 1.2], Standard Error of Mean 0.40
Statistical Analysis 2: Comparison: Placebo vs Tavapadon; Part II; Test type: Superiority; p = 0.0203, Mixed-effect Model Repeated Measurement — [p-value comment as in outcome 1, analysis 1]; LS Mean of Difference = -1.2, 95% CI 2-sided [-2.2 to -0.2], Standard Error of Mean 0.52
Statistical Analysis 3: Comparison: Placebo vs Tavapadon; Part III; Test type: Superiority; p = 0.0118, Mixed-effect Model Repeated Measurement — [p-value comment as in outcome 1, analysis 1]; LS Mean of Difference = -2.4, 95% CI 2-sided [-4.3 to -0.5], Standard Error of Mean 0.96

ADVERSE EVENTS:
Time Frame: All-cause mortality were reported from enrollment to the end of study, median time on follow up (median time subjects were followed) was 190 and 189 days for Placebo and Tavapadon, respectively. Treatment-emergent adverse events and serious adverse events were collected from first dose of study drug until 4 weeks after the last dose of study drug; mean duration on study drug was 169.6 and 151.7 days for Placebo and Tavapadon, respectively.
Arm/Group | Placebo | Tavapadon
All-Cause Mortality (participants affected / at risk) | 0/255 | 1/252
Serious Adverse Events (participants affected / at risk) | 14/255 | 17/252
Other Adverse Events (participants affected / at risk) | 90/255 | 130/252
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=255) | Tavapadon (N=252)
ANAEMIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
ANGINA PECTORIS (Cardiac disorders) | 0 (0) | 1 (1)
ATRIAL FIBRILLATION (Cardiac disorders) | 1 (1) | 0 (0)
CARDIAC FAILURE CHRONIC (Cardiac disorders) | 0 (0) | 1 (1)
GLAUCOMA (Eye disorders) | 0 (0) | 1 (1)
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 (0) | 2 (2)
DIARRHOEA (Gastrointestinal disorders) | 0 (0) | 1 (1)
HIATUS HERNIA (Gastrointestinal disorders) | 1 (1) | 0 (0)
BRONCHITIS BACTERIAL (Infections and infestations) | 0 (0) | 1 (1)
CELLULITIS (Infections and infestations) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 2 (2) | 0 (0)
COVID-19 PNEUMONIA (Infections and infestations) | 0 (0) | 1 (1)
EYE INFECTION (Infections and infestations) | 1 (1) | 0 (0)
INFECTIVE ANEURYSM (Infections and infestations) | 0 (0) | 1 (1)
LYME DISEASE (Infections and infestations) | 1 (1) | 0 (0)
SUBACUTE ENDOCARDITIS (Infections and infestations) | 0 (0) | 1 (1)
FALL (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
HIP FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
JOINT DISLOCATION (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
THERMAL BURN (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
HEPATIC ENZYME INCREASED (Investigations) | 0 (0) | 1 (1)
INTERVERTEBRAL DISC DISORDER (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
RHEUMATIC DISORDER (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
B-CELL SMALL LYMPHOCYTIC LYMPHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
PANCREATIC CARCINOMA METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
COLLOID BRAIN CYST (Nervous system disorders) | 1 (1) | 0 (0)
DIZZINESS (Nervous system disorders) | 0 (0) | 1 (1)
MIDDLE CEREBRAL ARTERY STROKE (Nervous system disorders) | 0 (0) | 1 (1)
ON AND OFF PHENOMENON (Nervous system disorders) | 1 (1) | 0 (0)
SUBARACHNOID HAEMORRHAGE (Nervous system disorders) | 0 (0) | 1 (1)
ANXIETY DISORDER (Psychiatric disorders) | 1 (1) | 0 (0)
HALLUCINATION, VISUAL (Psychiatric disorders) | 0 (0) | 1 (1)
SUICIDAL IDEATION (Psychiatric disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=255) | Tavapadon (N=252)
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 (1) | 6 (6)
CONSTIPATION (Gastrointestinal disorders) | 8 (9) | 10 (10)
DRY MOUTH (Gastrointestinal disorders) | 2 (2) | 7 (7)
NAUSEA (Gastrointestinal disorders) | 11 (14) | 36 (44)
ASTHENIA (General disorders) | 0 (0) | 8 (8)
FATIGUE (General disorders) | 11 (11) | 10 (11)
COVID-19 (Infections and infestations) | 7 (7) | 13 (13)
NASOPHARYNGITIS (Infections and infestations) | 6 (6) | 7 (7)
URINARY TRACT INFECTION (Infections and infestations) | 7 (9) | 7 (10)
CONTUSION (Injury, poisoning and procedural complications) | 6 (7) | 4 (4)
FALL (Injury, poisoning and procedural complications) | 13 (20) | 13 (18)
WEIGHT DECREASED (Investigations) | 1 (1) | 7 (7)
DECREASED APPETITE (Metabolism and nutrition disorders) | 1 (1) | 6 (6)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 7 (7) | 5 (5)
DIZZINESS (Nervous system disorders) | 8 (8) | 18 (20)
DYSGEUSIA (Nervous system disorders) | 0 (0) | 7 (7)
DYSKINESIA (Nervous system disorders) | 4 (7) | 25 (32)
DYSTONIA (Nervous system disorders) | 0 (0) | 7 (9)
HEADACHE (Nervous system disorders) | 7 (7) | 17 (23)
SOMNOLENCE (Nervous system disorders) | 11 (11) | 13 (13)
ANXIETY (Psychiatric disorders) | 7 (7) | 8 (8)
DEPRESSION (Psychiatric disorders) | 2 (2) | 6 (7)
HALLUCINATION, VISUAL (Psychiatric disorders) | 3 (3) | 13 (14)
INSOMNIA (Psychiatric disorders) | 7 (7) | 1 (1)
HYPERHIDROSIS (Skin and subcutaneous tissue disorders) | 6 (6) | 3 (3)
HYPOTENSION (Vascular disorders) | 1 (1) | 9 (9)
ORTHOSTATIC HYPOTENSION (Vascular disorders) | 3 (3) | 15 (15)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2023-07-06): https://cdn.clinicaltrials.gov/large-docs/99/NCT04542499/Prot_000.pdf
  • Statistical Analysis Plan (2024-03-11): https://cdn.clinicaltrials.gov/large-docs/99/NCT04542499/SAP_001.pdf